CLINICAL TRIAL: NCT06299514
Title: Resynchronization for Ambulatory Heart Failure Trial in Patients With Chronic Atrial Fibrillation - Pharmacological Rate Control vs. Pace and Ablate With Conduction System Pacing
Brief Title: RAFT - Pace &Ablate
Acronym: RAFT-P&A RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Habib Khan (Other)
Responsible Party: Sponsor-Investigator, Habib Khan, Cardiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4754
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Heart Failure; Pacemaker; Arrhythmia Atrial
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacological Therapy (Active Comparator): Patients randomized to pharmacology rate control will receive guideline-directed HF management across all ranges of LVEF, including appropriate rate control medications. ICD will be inserted in those patients who have LVEF ≤35%
  Interventions: Drug: Medication
- P&A-CSP (Experimental): Patients randomized to P&A-CSP will receive a CSP and ICD if LVEF ≤35% within 10 working days of randomization. Catheter AVNA will be performed within 4 weeks.
  Interventions: Device: Pace and Ablate

INTERVENTIONS:
Device: Pace and Ablate — Conduction System Pacing (CSP) followed by AtrioVentricular Node Ablation (AVNA)
  Other Names: P&A, pacemaker and atrioventricular node ablation
  Arms: P&A-CSP
Drug: Medication — Optimization of heart failure therapies includes maximum tolerated doses of beta-blockers, aldosterone antagonists, ACE inhibitors, ARB, diuretics, ARNis
  Other Names: Optimal heart failure therapy
  Arms: Pharmacological Therapy

SUMMARY:
Atrial fibrillation (AF) is an irregular heartbeat that can cause symptoms of skipped beats, shortness of breath, stroke, or in some cases fluid in the lungs or legs. Treating AF is mostly to do with slowing the heart rate down so that the heart can get a chance to regain some energy. In some cases, slowing the heart rate is not easy to achieve as some patients find it difficult to tolerate medications and suffer side effects from these treatments. In these instances, there might be a possibility to permanently control the heart rate by implanting a pacemaker in the heart and intentionally damaging a regulatory region of the heart called the atrioventricular (AV) node. Damaging the AV node by a procedure called ablation results in the AF not being able to influence the bottom chambers (the ventricles) resulting in a slow rhythm. Therefore, if a pacemaker is implanted then the heart rate can be completely regulated by the pacemaker.

A complex pacemaker that stimulates both the right and left ventricles simultaneously (BiVP) has been used for the last decade prior to AV node ablation. More recently, a technique has been designed to reduce the number of leads in the heart, reduce procedure time and have a similar effect on the heart called Conduction System Pacing (CSP). There is not enough existing evidence to show that a pace and ablate strategy is superior to optimal medical therapy. We intend to compare the efficacy of CSP with AV node ablation to optimal medical therapy for treating AF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with permanent AF/persistent AF (in AF)
2. Patients with NYHA Class II -IVa HF symptoms
3. Guideline driven medical therapy for HF for at least 3- months with an NT-proBNP ≥ 900 ng/L, or ≥ 600 ng/L if the patient has had a HF hospitalization within 1 year

Exclusion Criteria:

1. In hospital patients needing intensive care or intravenous inotropic agent in the last 4 days
2. Patients with a life expectancy of ≤ 1 year from non-cardiac cause or anticipating a transplant within 1 year
3. Acute coronary syndrome <4 weeks or coronary revascularization <3months
4. Unable or unwilling to provide informed consent
5. Uncorrected primary valvular disease or prosthetic tricuspid valve
6. Restrictive, hypertrophic, or irreversible form of cardiomyopathy
7. Severe pulmonary diseases requiring oxygenation
8. Patients with a known history of WHO Class I pulmonary hypertension (PH) which includes PH associated with CVD, collagen vascular disease, congenital shunts, cirrhosis and portal hypertension, HIV, hemoglobinopathies, schistosomiasis or drug-associated PH as well as those with high suspicion of irreversible pulmonary hypertension
9. Patients enrolled in competitive clinical trials that will affect the objectives of this study
10. Existing CRT/BiVP
11. Patients who are pregnant
12. Guideline indication for CRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Winratio | 12 months
  Reduction in the hierarchical composite outcomes of all-cause mortality and HF events frequency, improvement in NT-proBNP and improvement in QOL.

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  Mortality from any cause within the 12 month of follow up period
Cardiovascular mortality | 12 months
  Mortality attributed to cardiovascular causes within 12 month follow up period
Number of heart failure events | 12 months
  Heart failure related presentations to health care facilities necessitating intravenous diuretics or overnight stay
All-cause hospitalization | 12 months
  ER admission or overnight stay
Quality of Life -Kansas City Cardiomyopathy Questionairre (KCCQ) | 6 months
  Change in Kansas HF score from baseline. KCCQ is a 23-item self-administered questionnaire that measures the participant's perception of their health status, including their HF symptoms, impact on physical and social function and how their HF impacts the quality of life (QoL). KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), QoL (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status.
Exercise | 6 months
  Change in 6 minute walk distance from baseline
Biochemical marker | 6 months
  Change in NTproBNP from baseline
Cognitive assessment | 12 months
  Change in cognitive assessment scores from baseline

CONTACTS AND LOCATIONS:
Locations (12):
- Canada (12):
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Waterloo Wellington Cardiovascular Research Institute, Kitchener, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Ottawa Heart Institute Research Corporation, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier de L'Université de Montréal (CHUM), Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie Québec - Université Laval (IUCPQ-ULaval), Québec, Quebec
  - Hôpital Fleurimont, Sherbrooke, Quebec